CLINICAL TRIAL: NCT03969147
Title: Investigation of a Novel Oropharyngeal Airway: The ManMaxAirway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kalev Freeman, Assistant Professor of Surgery, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS 16-105
Record Dates: First submitted 2018-02-16; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Airway Obstruction; Respiratory Complication
MeSH Terms: conditions — Airway Obstruction

ARMS (3):
- MRI Comparison (Active Comparator): MRI images will be obtained of the airways of healthy volunteers both with the ManMaxAirway oropharyngeal airway adjunct and with no airway adjunct in place in order to observe any changes to the airway anatomy caused by placement of the airway adjunct. The order of the scans (with and without airway adjunct) will be determined by randomization software in advance.
  Interventions: Device: ManMaxAirway oropharyngeal airway adjunct; Device: No airway adjunct
- Tolerability Comparison (Experimental): Healthy volunteers will self-place either the ManMaxAirway oropharyngeal airway adjunct or the Guedel Oropharyngeal airway adjunct, which will be left in place for an interval of one minute, while supervised by research staff. After completing a questionnaire and resting for a timed interval, they will then self-place the other airway adjunct, which will be left in place for the same length of time as the first, before completing another questionnaire. The order in which the devices are placed by each subject will be determined in advance via computer randomization.
  Interventions: Device: ManMaxAirway oropharyngeal airway adjunct; Device: Guedel Oropharyngeal airway adjunct
- Forced Oscillation (Active Comparator): Volunteers from the tolerability comparison arm will also be invited as a subset of subjects to participate in a measurement of resistance to forced oscillation. The volunteers will be subject to forced oscillations in a pulmonary function lab with the ManMaxAirway oropharyngeal airway adjunct in place and with no airway adjunct in order to observe changes in resistance to oscillatory airflow
  Interventions: Device: ManMaxAirway oropharyngeal airway adjunct; Device: No airway adjunct

INTERVENTIONS:
Device: ManMaxAirway oropharyngeal airway adjunct — Healthy volunteers will self-place the ManMaxAirway.
Device: Guedel Oropharyngeal airway adjunct — Healthy volunteers will self-place the standard Guedel OPA.
  Arms: Tolerability Comparison
Device: No airway adjunct — Healthy volunteers will have no airway adjunct in place.
  Arms: Forced Oscillation; MRI Comparison

SUMMARY:
Guedel pattern or oropharyngeal airways (OPA) maintain an open oral airway in unconscious or semi-conscious patients by preventing the tongue from covering the epiglottis, but OPA placement carries a risk of inducing gag reflex and vomiting. Although various sizes are available, the design of the OPA has undergone little change since its introduction in the 1920s. The purpose of this study is to determine the utility of a novel airway device, the ManMaxAirway (MMA), as an alternative to the OPA.

DETAILED DESCRIPTION:
Oropharyngeal airways are simple devices placed in the mouth that help to maintain an open oral airway in anesthetized or otherwise unconscious or semi-conscious patients and also help to facilitate assisted ventilation with a bag and mask. The current standard of care, the Guedel airway, was originally designed by Dr. Arthur Guedel in 1933 and has remained essentially unchanged since its inception. It is a narrow, curved plastic tube which slides over the tongue to lie in the back of the throat. While this device has withstood the test of time, proving to be largely safe and effective, it is known to have several drawbacks: 1) it is not held securely in place in the mouth which allows it to become easily mal-positioned or expelled, 2) it often triggers a gag reflex in even minimally conscious patients limiting its utility in emergency and prehospital settings, 3) there are case reports of serious complication and injury as a result of the poor fit and retention of the Guedel airway including aspiration and injury to the tongue, posterior pharynx, and teeth, and 4) the Guedel airway's narrow and rigid construction make it unsuitable for patients who may clench their teeth, such as in patients who are seizing.

The purpose of this study is to obtain preliminary data to help determine the utility of the ManMaxAirway (MMA) for ventilation and that will aid in future study designs for the device. The MMA is a novel oral airway that is similar in size and shape to an athletic mouth guard, and which fits between and is held in place by the teeth (or gums of the edentulous patient). The external portion of the airway contains a flange in the front which remains anterior to the teeth, allowing for ventilation in a similar fashion to the Guedel airway. It also has a central lumen that divides posterior to the flange into two lateral passages, such that air passes through the U-shaped device to the posterior-lateral aspect of the tongue behind the back teeth. Unlike the Guedel device, it makes little contact with the tongue and does not protrude into the posterior pharynx. Instead, the device will - in theory - force the mandible to rest slightly anterior to the maxilla: this slight mandible-maxilla displacement (similar to that achieved via the jaw thrust technique) will theoretically allow for a better opening of the airway without requiring direct depression of the tongue. We hypothesize that the ManMaxAirway will maintain a viable airway and allow for adequate ventilation of patients while demonstrating the following advantages over the Guedel airway: 1) improved tolerability and ease of insertion with decreased gag reflex stimulation in conscious patients 2) ability to act as a bite block in patients actively seizing or likely to seize.

Our proposed study will include two major aims in assessing the utility of the MMA. Our first aim will be to assess the mechanical effect of the device on the oropharyngeal anatomy. We will obtain MRI images of several healthy volunteers, with and without the MMA in place, in order to observe any displacement of the mandible relative to the maxilla, and any changes in positioning of the tongue. We will also assess the physical performance characteristics of the MMA vs. Guedel in terms of flow resistance in the simulation laboratory. Our second aim will be to determine whether there is any difference in tolerability between the Man Max Airway and the Guedel airway. To address the second aim we propose a crossover study using conscious, healthy volunteers, in which subjects will be asked to place each device in their mouth, one after the other. We will document the elapsed time and the number of breaths that subjects are able to take with each device in place (up to one minute), and will obtain ratings of device discomfort from each subject using a visual analog scale. We will also measure resistance to forced oscillatory airflow in a subset of subjects, with and without the airway in place, at a second visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over the age of 18.

Exclusion Criteria:

* For Tolerability arm: History of Gastroesophageal Reflux Disease, dental implants or dental prostheses
* For the MRI arm, the following were further exclusion criteria as dictated by institutional MRI safety protocols: claustrophobia, cerebral aneurysm clip, nerve stimulation device, cochlear/middle ear implant, transdermal patches, known metal in body (to include IUD), intraventricular shunt, implanted pumps or stents, pregnant, metal implants, cardiac pacemaker, Swan Ganz catheter, metal worker occupation, history of eye injury with metal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability to place the Novel Airway Adjunct | 1 minute (During tolerability comparison experiment)
  Any inability of conscious, healthy volunteers to place the device (MMA) in their mouth will be recorded.

SECONDARY OUTCOMES:
Displacement of the mandibular condyle and the condylar fossa apex (MRI arm) | 2-3 weeks following MRI scans.
  A radiologist will measure displacement (mm) between the mandibular condyle and condylar fossa apex using MRI on healthy subjects with and without the device (MMA) in place.
Number of respirations with airway adjunct in place (Tolerability Arm) | 1 minute (During tolerability comparison experiment)
  Recorded by research staff while healthy subject has airway adjunct (either MMA or OPA) in place.
Elapsed time (up to 60 seconds) that subject is able to tolerate having the airway adjunct in place (Tolerability Arm) | 1 minute (During tolerability comparison experiment.)
  Recorded by research staff while healthy subject has airway adjunct (either MMA or OPA) in place.
Visual Analog Tolerability | 1 minute (following tolerability comparison experiment.)
  100 mm line that subjects will use to mark level of discomfort for each device (MMA or OPA), with 0mm correlating to complete tolerability with no discomfort and 100mm correlating to completely intolerable discomfort.
Resistance to oscillatory air flow | 1 minute (Assessment done following physical lab tests)
  Airflow resistance (cmH20·s/L) of the two devices (MMA and OPA) will be compared using forced oscillations measured in a pulmonary lab.

CONTACTS AND LOCATIONS:
Overall Officials: Kalev Freeman, MD, PhD, Principal Investigator — University of Vermont Department of Surgery
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No